CLINICAL TRIAL: NCT07267611
Title: Evaluating the Reliability and Validity of the Arabic Version of the SAMANTA Questionnaire: A Step Toward Improved Diagnosis of Heavy Menstrual Bleeding.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Abdel Raheem, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: SAMANTA HMB
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: Reproductive age women, from 15 to 45 years old with heavy Menstrual Bleeding.

SUMMARY:
Heavy menstrual bleeding (HMB) significantly impacts women's quality of life (QoL). However, despite the high prevalence of HMB, culturally adapted screening tools remain scarce in our locality. This study aimed to adapt and validate the Arabic version of SAMANTA questionnaire for non-pregnant women of reproductive age.

HMB can primarily be a consequence of structural or functional disturbances within the reproductive system, but it may also be linked to structural and functional ailments of other bodily systems (vascular abnormalities, malignancies, or coagulation disorders) With the exact global prevalence varies from 4% to 51% across different countries and racial groups, with estimates suggesting that approximately one-third of reproductive-age women experiences HMB .

HMB is deﬁned as excessive menstrual blood loss which interferes with a woman's physical, social, emotional and/or material quality of life. It can occur alone or in combination with other symptoms. The term heavy menstrual bleeding has replaced the term menorrhagia.

The gold standard for the measurement of blood in sanitary products is the extraction of hematin using a 5% sodium hydroxide solution and the estimation of the alkaline hematin content by spectrophotometry .

This method is not feasible in clinical practice and has only been used in research studies.

HMB can cause iron-deficiency anemia, which is among the leading causes of years lived with disability in low-income and middle-income countries (LMICs). It is also associated with a range of adverse functional outcomes, including lower productivity and income earning, reduced ability to perform daily activities, and limitations on social life and relationships.

Recent research in the area of HMB has recognized the importance of measuring "patient experience" as an outcome and the National Institute of Clinical Excellence from the UK suggests that any intervention for HMB should aim to improve quality of life rather than focusing on menstrual blood loss .

For women with HMB early and accurate diagnosis is important to prevent its negative consequences. However, in low resource settings, facilities are not always available. For this reason, a cheap, simple to use tool to identify women with HMB and its impact on their quality of life is needed.

In the present study, we test the ability of the Arabic version of SAMANTA-Q as a simple tool to identify women with HMB.

ELIGIBILITY:
Inclusion Criteria:

* women, from 15 to 45 years old
* Reproductive age women

Exclusion Criteria:

Women with amenorrhea. Postmenopausal women. Pregnant women. Women who had given birth within the previous 6 months. Women with mental illness, or inability to make decisions or follow instructions.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Reproductive age women, from 15 to 45 years old were eligible for the study
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
accuracy of Arabic Version of the SAMANTA Questionnaire | baseline